CLINICAL TRIAL: NCT00708331
Title: SC25-FOLD Hydrophilic Acrylic Intraocular Lens
Brief Title: Hydrophilic Acrylic Intraocular Lens
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: EyeKon Medical, Inc. (Industry)
Responsible Party: Mark D. Robinson, President and CEO, EyeKon Medical, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EyeKon SC25-FOLD
Record Dates: First submitted 2008-06-30; First posted 2008-07-02 (Estimated); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Cataract Extraction
Keywords: Cataract; Extraction; Intraocular Lens; Hydrophilic Acrylic
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Device: 2 HEMA Hydrophilic Acrylic Intraocular Lens

INTERVENTIONS:
Device: 2 HEMA Hydrophilic Acrylic Intraocular Lens — 2 HEMA Hydrophilic Acrylic Intraocular Lens implanted into the posterior capsule following cataract surgery for patient life duration.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Hydrophilic Acrylic Intraocular Lens after cataract surgery

ELIGIBILITY:
Inclusion Criteria:

* The patient is in good general and ocular health, having a vision-reducing cataract in the intended operative eye
* The patient is willing and able to complete all required postoperative visits.
* The patient is willing to sign a statement of informed consent.

Preoperative Exclusion Criteria:

* The patient is under the age of 18
* The patient has had prior intraocular surgery in the operative eye.
* The patient has systemic diseases with ocular manifestations (e.g. diabetes, complications of immune deficiency syndrome), which may contribute to postoperative confounding of data interpretation.
* The patient's worst seeing eye is 20/70 or worse.
* The patient has multiple surgical procedures at the time of implant.
* The patient has chronic use of steroids, immunosuppressive and/or antineoplastic agents.
* The patient has acute infection, inflammation of the eye.
* Iris atrophy
* Proliferative diabetic retinopathy.
* Chronic, medically uncontrolled glaucoma
* Chronic uveitis, iritis, iridocyclitis or rubeosis of the lids
* Rubella, traumatic or congenital/developmental cataract.
* Severe retinal pathology (e.g. retinal tear, detachment, etc).

Operative Patient Exclusion Criteria

* Capsular rupture
* Vitreous loss
* Hyphema
* Zonular disinsertion
* Surgical Complications- In the event of a complication during surgery, the surgeon should decide whether the stability of the hydrophilic acrylic lens would be compromised by the complication, e.g. in the event of zonular damage of major capsule rupture. If the lens stability would be compromised, the hydrophilic acrylic lens should not be implanted and the surgeon should make arrangements to implant an alternative lens.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2002-08; Primary Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Visual Acuity | At all pre/post op CRFs for 2 yrs

SECONDARY OUTCOMES:
Adverse Events | 2yrs

CONTACTS AND LOCATIONS:
Overall Officials: James Garvey, M.D., Study Director; David C Brown, M.D., Principal Investigator — Eye Centers of Florida; Michael S Korenfeld, M.D., Principal Investigator — Comprehensive Eye Care LTD; James E Croley, M.D., Principal Investigator — Cataract and Refractive Institute of Florida; Larry Perich, D.O., Principal Investigator — The Perch Eye Center; Thomas L Croley, M.D., Principal Investigator — Central Florida Eye Institute; Farrell C Tyson, M.D, Principal Investigator — Cape Coral Eye Center; James P Gills, M.D., Principal Investigator — St. Lukes Cataract and Laser Center; Robert Weinstock, M.D, Principal Investigator — The Eye Institute of West Florida
Locations (9):
- United States (9):
  - Cape Coral Eye Center, Cape Coral, Florida
  - Cataract and Refractive Institute of Florida, Cape Coral, Florida
  - Eye Centers of Florida, Fort Myers, Florida
  - Riverside Park Surgicenter, Jacksonville, Florida
  - The Eye Institute of West Florida, Largo, Florida
  - The Perich Eye Center, New Port Richey, Florida
  - Central Florida Eye Institute, Ocala, Florida
  - St. Lukes Cataract and Laser Center, Tarpon Springs, Florida
  - Comprehensive Eye Care Ltd., Washington, Missouri